CLINICAL TRIAL: NCT06082089
Title: A Structured and Empirically Validated Multidimensional Intervention Program to Improve Postdivorce Adjustment and Psychological Well-Being for Divorced Women
Brief Title: Divorce Adjustment Program for Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Adviye Esin Yılmaz, Professor, Clinical Psychologist, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 218K458
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Divorced; Adjustment Reaction
Keywords: divorce; postdivorce adjustment; psychological well-being; intervention program
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postdivorce Intervention Program (Experimental): The experimental arm will receive the 5- or 6-session online group intervention program developed for divorced women.
  Interventions: Behavioral: Divorce Adjustment Program (DAP)
- Wait List and Delayed Intervention (No Intervention): In this arm, participants in the wait list control group will complete outcome measures without the intervention program being implemented. After the post intervention assessments are completed, this group will receive either the online intervention program or booklets including detailed information about the program, depending on their preference.

INTERVENTIONS:
Behavioral: Divorce Adjustment Program (DAP) — This is a brief group intervention program for divorced women. It consists of 6 sessions for participants with children and 5 sessions for participants without children. Each session lasts approximately 2.5-3 hours focusing on one of the difficulties experienced by women after divorce (i.e., self-perception, emotions and emotion regulation, social problems, family-related problems, problems with ex-spouse and children (for participants with children)). In this study, the DAP will be implemented in online format.
  Arms: Postdivorce Intervention Program

SUMMARY:
This study is the randomized controlled trial (RCT) part of a broader project aiming to develop and evaluate the effectiveness and feasibility of a structured, culture-sensitive brief divorce adjustment program (DAP) for women. The present pilot RCT will be the first to test the potential effectiveness of the DAP to be delivered in an online group format in comparison to a wait-list control group. The feasibility of the program will be evaluated considering the percentages of attendance to the sessions, drop-out rates and qualitative assessments at the end of each session, as well as at the end of the program.

DETAILED DESCRIPTION:
Considering the current pattern of rising divorce rates in all over the world, multi-dimensional, culturally-sensitive and well-structured interventions available for people in the post-divorce period has crucial importance in clinical practice. The divorce adjustment program (DAP) is such an group intervention that is designed in the previous stage of this study to improve the level of postdivorce adjustment and psychological well-being.

The main purpose of this study is to test the potential effectiveness of the DAP to be delivered in an online group format for Turkish women who might undergo a more challenging adaptation process than that of men as indicated by the relevant literature. The DAP is a 5-module intervention for women without children and has an extra children-focused module, making the program 6 modules for women with children.

Since the DAP has not been used and/or tested before, this study will be designed as a pilot RCT in which the program will be implemented in an online group format to Turkish divorced women reporting adjustment difficulties (as determined by having scores on the Fisher Divorce Adjustment Scale-Short Form [FDAS-SF] below the average that of reported in the Turkish adaptation study). The potential effectiveness of the DAP will be tested compared to a wait-list control group (with delayed intervention). On taking baseline assessments, eligible 60 participants with children and 60 participants without children will separately be randomized to either the experimental DAP group (n = 30 for women with children; n = 30 for women without children) or to the wait-list control group (n = 30 for women with children; n = 30 for women without children). If the time gap between baseline assessment and the first DAP session exceeds 1-week period, the pre-intervention assessments will be recurred. The effectiveness of the program will be evaluated by means of various measurements to be taken before the intervention, immediately after the completion of the program and at 1-month and 3-month follow-ups. All divorced women including drop-outs will be invited to outcome assessments. After completion of the follow-up assessment, the wait-list participants will be given opportunity to choose either participation to the DAP or receiving booklets including detailed information about the DAP content. The primary outcome measure will be divorce adjustment score and depression, anxiety, stress, life satisfaction, psychological well-being, and ego strength measures will be the secondary outcomes.

The feasibility of the program will be evaluated by assessing the percentages of attendance to the sessions, drop-out rates and qualitative assessments at the end of each session, as well as at the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Being legally divorced
* Adjustment difficulties to divorce as indicated by having a FDAS-SF score of 98 or below for those with children and 94 or below for those without children (these scores are the average scores determined in the FDAS-SF Turkish adaptation study)
* Not being remarried or involved in a current romantic relationship
* Not receiving concurrent psychotherapy

Exclusion Criteria (as determined by the Diagnostic and Statistical Manual-5 [DSM-5] Level 1 Cross-Cutting Symptom Measure and a confirmatory telephone screening with the eligible participants):

* Substance use problems
* Suicidal thoughts
* Psychotic symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Fisher Divorce Adjustment Scale-Short Form (FDAS-SF) | Change from baseline assessment, at 1 week post-intervention assessment (6-7 weeks after baseline), change from post-assessment at 1 month post-intervention assessment (2.5-3 months after baseline), and change from at 3 month post intervention assessment
  The FDAS-SF is a 25-item measure of postdivorce adjustment in terms of grief reactions, disentanglement from the relationship, anger, trust and intimacy, and self-worth. Items are scored as 5 (always) to 1 (never), providing a range between 25 to 125. Higher scores indicate higher levels of adjustment to divorce.

SECONDARY OUTCOMES:
The Depression Anxiety Stress Scale-21 (DASS-21) | Change from baseline assessment, at 1 week post-intervention assessment (6-7 weeks after baseline), change from post-assessment at 1 month post-intervention assessment (2.5-3 months after baseline), and change from at 3 month post intervention assessment
  It is a 21-item psychological distress measure assessing the presence and severity of symptoms of depression, anxiety and stress as separate components. The items are rated on a 4-point scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much, or most of the time). Since the DAS-21 is a shorter version of the 42 item DASS, the scores should be multiplied by 2 for calculating the final score of the DASS-21 subscales. The ratings can be classified as normal, mild, moderate, severe, and extremely severe.
The Satisfaction With Life Scale (SWLS) | Change from baseline assessment, at 1 week post-intervention assessment (6-7 weeks after baseline), change from post-assessment at 1 month post-intervention assessment (2.5-3 months after baseline), and change from at 3 month post intervention assessment
  The SWLS is a 5-item measure of an individual's judgment of satisfaction with life as a whole. The items scored on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree), revealing a range between 5 to 35. Higher scores indicate higher levels of life satisfaction.
Psychological Well-Being Scale (PWBS) | Change from baseline assessment, at 1 week post-intervention assessment (6-7 weeks after baseline), change from post-assessment at 1 month post-intervention assessment (2.5-3 months after baseline), and change from at 3 month post intervention assessment
  The PWBS is a 8-item scale developed to evaluate socio-psychological well-being. Items are scored on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). The total score of the PWBS ranges between 8 to 56 and higher scores indicate higher levels of psychological well-being.
The Ego-Resiliency Scale (ERS) | Change from baseline assessment, at 1 week post-intervention assessment (6-7 weeks after baseline), change from post-assessment at 1 month post-intervention assessment (2.5-3 months after baseline), and change from at 3 month post intervention assessment
  It is a 14-item scale that aims to assess the ability to adapt to stress and adversity. Items are scored on a 4-point Likert-scale ranging from 1 (Does not apply at all) to 4 (Applies very strongly). Higher scores indicate higher levels of psychological resilience.